CLINICAL TRIAL: NCT04139460
Title: CRT-P or CRT-D in Patients With Dilated Cardiomyopathy and Heart Failure Without LGE-CMR High-risk Markers
Brief Title: CRT-P or CRT-D in Dilated Cardiomyopathy
Acronym: CRT-REALITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Tomas Skala, MD, PhD, FESC, Principal investigator, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University Hospital Olomouc
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiomyopathy, Dilated, 3B
Keywords: Non-ischemic cardiomyopathy; Heart failure; Implantable cardioverter-defibrillator; Cardiac resynchronization therapy; Magnetic resonance imaging; Late gadolinium enhancement
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, interventional parallel-design trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial participants will be blinded to the device type for the whole duration of the trial.
  The randomizing and implanting physicians will not be blinded to the type of the device. These physicians will not take care in the subsequent patients' follow-up and sign a declaration of confidentiality.
  The same will be true for the physicians / technicians attending to the device interrogation during follow-up visits. The device type will be hidden and physicians will sign a declaration of confidentiality. The patients' documentation will not reveal the device type.
  A maximum effort will be done to hide the type of the implanted device. The implantation will be intramuscular and the device interrogation follow-up visits will not reveal the device type.
  The physicians attending the follow-up visits and entering all patients' data into web-based CRF will be blinded to the implanted device type.
  The outcomes assessors will also be blinded to the implanted device type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT-D (Active Comparator): Implantation of cardiac resynchronization therapy with a defibrillator (CRT-D)
  Interventions: Device: CRT-D
- CRT-P (Active Comparator): Implantation of cardiac resynchronization therapy pacemaker (CRT-P)
  Interventions: Device: CRT-P

INTERVENTIONS:
Device: CRT-D — After randomization, devices will be implanted as soon as possible (within 2 weeks). The ICD will be programmed with anti-tachycardia pacing and shock therapy as per common praxis.
  Arms: CRT-D
Device: CRT-P — After randomization, devices will be implanted as soon as possible (within 2 weeks).
  Arms: CRT-P

SUMMARY:
The ICD-Reality study is a non-commercial, investigator-led, multicenter, prospective, randomized, controlled trial. We aim to determine the effect of CRT-D or CRT-P implantation in non-ischemic cardiomyopathy and heart failure patients.

The reason why we initiated this trial is the lack of evidence-based treatment for the significant number of these patients. In these patients, 5-year mortality remains as high as 20% despite recent therapeutic advances. Based on currently available evidence, because of a significant decrease in mortality due to modern pharmacotherapy, it is not certain which of these patients should receive a CRT-P and who should receive a CRT-D. No dedicated and adequately powered trial has addressed this important question.

We hypothesize that patients with symptomatic HF, LVEF ≤35%, without left ventricular mid-wall fibrosis on LGE-CMR, will not benefit from CRT-D implantation compared with CRT-P only implantation.

If our hypothesis is confirmed, this could provide evidence for the management of these patients with a significant impact on common daily praxis and health care expenditures.

We aim to enroll 600 patients in the trial. 924 patients are needed to be screened for these 600 patients to be randomized.

Patients with non-ischemic HF visiting an out-patient department and possibly eligible for the trial will have their pharmacotherapy optimized.

Patients with a significant amount of fibrosis will be excluded from the study and treated according to local practice with an emphasis on ICD implantation to prevent SCD.

After fulfilling all eligibility criteria, including maximally tolerated pharmacotherapy, subjects will be randomized by the physicians who enrolled them in a 1:1 ratio to receive CRT-D or CRT-P implantation.

All patients will be followed-up for at least 3 years after the implantation.

DETAILED DESCRIPTION:
The trial goals The ICD-Reality study is an investigator-led, multicenter, prospective, randomized, controlled trial. We aim to determine the effect of CRT-D or CRT-P implantation in non-ischemic cardiomyopathy and heart failure patients. The reason why we initiated this trial is the lack of evidence-based treatment for the significant number of these patients. In these patients, 5-year mortality remains as high as 20% despite recent therapeutic advances. Based on currently available evidence, because of a significant decrease in mortality due to modern pharmacotherapy, it is not certain which of these patients should receive an ICD. We hypothesize that patients with symptomatic HF, LVEF ≤35%, without left ventricular mid-wall fibrosis on LGE-CMR, will not benefit from CRT-D implantation compared with CRT-P only implantation. If our hypothesis is confirmed, this could provide evidence for the management of these patients with a significant impact on common daily praxis and health care expenditures.

Clinical hypothesis:

Patients with symptomatic HF, with LVEF ≤35% and without LV mid-wall fibrosis on late gadolinium enhancement cardiovascular magnetic resonance imaging (CMR), will not benefit from CRT-D implantation compared with CRT-P only implantation.

Estimated number of patients needed to be screened and randomized:

600 patients are needed to be randomized according to the study power analysis. Since 35 % of patients are estimated to be LG-E positive and thus excluded from randomization, 924 patients are needed to be screened.

Pre-screening:

Patients with non-ischemic HF visiting an out-patient department and possibly eligible for the trial will have their pharmacotherapy optimized. A screening visit in an out-patient department will be scheduled in 1-2 months after pharmacotherapy optimization since the qualifying LVEF and NT-proBNP level has to be measured after a maximal tolerated pharmacotherapy of heart failure has been achieved.

Screening:

After the signing of informed consent, screening examination will be performed. The informed consent will be obtained by attending physician in every center and a signed original will be stored in each individual center for the whole duration of the study. The screening examination will include medical history, documentation of underlying cardiac disease. The following co-morbidities will be specifically documented: peripheral arterial disease, cerebral vascular disease, pulmonary disease, diabetes mellitus, hypertension, sleep apnea, tobacco use, and any malignant disease within the last 5 years. Physical exam with vital signs, NYHA functional class, pulse rate, resting blood pressure will be performed. Cardiovascular pharmacological treatment will be documented. Standard laboratory parameters are recorded, including creatinine, estimated glomerular filtration rate, liver tests, TSH, NT-proBNP. Transthoracic echocardiography will be done to confirm LVEF ≤35% using biplane Simpson's method. Documented will be LV end-systolic and end-diastolic diameters and volumes, thickness of ventricular septum and LV posterior wall, stroke volume, cardiac output, indexed left atrial volume, presence and grade of valvular heart disease, right ventricle diameter, TAPSE, presence and grade of pulmonary hypertension. Selective coronarography will be performed if it was not done before to exclude patients with a severe coronary heart disease. LGE-CMR imaging will be performed by an operator blinded to all other clinical data to evaluate left ventricular mid-wall fibrosis.

Patients with a significant amount of fibrosis will be excluded from the study and treated according to local practice with an emphasis on ICD implantation to prevent SCD.

Randomization:

After fulfilling all eligibility criteria, including maximally tolerated pharmacotherapy, subjects will be randomized by the physicians who enrolled them in a 1:1 ratio to receive CRT-D or CRT-P implantation. Randomization will be carried out by physicians enrolling patients through a stand-alone web-based CRF managed by an independent biomedicine and statistics center, independent on all randomizing personnel. The web-CRF-based allocation sequence will be based on computer-generated random numbers and will be concealed until the type of intervention is assigned.

Treatment:

After randomization, devices will be implanted as soon as possible (within 2 weeks). The ICD will be programmed with anti-tachycardia pacing and shock therapy as per common praxis.

Follow-up:

All patients will be followed-up for at least 3 years after the implantation. After the implantation, all patients will be examined every 6 months in an out-patient department with the assessment of medical history, vital signs, physical exam, and NT-proBNP as in the screening visit. A device control will be performed every 6 months.

After device implantation the concomitant care and all possible concomitant interventions will be carried out as per common praxis.

Patients will be evaluated for possible end-points. Deaths and hospitalizations for heart failure, stroke or arrhythmias will be recorded throughout the study duration.

Quality of life (QoL) is assessed at baseline and annually during follow-up. Patients will fill out the SF-36 Questionnaire for general QoL, the MacNew Questionnaire for disease specific QoL.

An Endpoint Classification Committee will adjudicate hospitalizations and deaths for causality. An independent Data Monitoring Committee will periodically review mortality data throughout the study.

For safety reasons, all patients will be followed using a daily ECG monitoring and analysis. ECG from the Home-monitoring units will be evaluated in a dedicated center. This center will evaluate the ECGs sent from the Home-monitoring units with respect to patient safety and the study end-points. If the Home-monitoring unit reveals any rhythm disturbance they will contact the patient's physician and make a record in the CRF. If a sustained ventricular tachyarrhythmia is documented on a Home-monitoring in a CRT-P patient, a decision will be made and documented about a possible crossover to CRT-D as soon as possible.

Patients who will deviate from intervention protocols (e.g. crossover to CRT-D implantation) will continue to be followed-up.

Blinding:

Trial participants will be blinded to the device type for the whole duration of the trial.

The randomizing and implanting physicians will not be blinded to the type of the device. These physicians will not take care in the subsequent patients' follow-up and sign a declaration of confidentiality.

The same will be true for the physicians / technicians attending to the device interrogation during follow-up visits. The device type will be hidden and physicians will sign a declaration of confidentiality. The patients' documentation will not reveal the device type.

A maximum effort will be done to hide the type of the implanted device. The implantation will be intramuscular and the device interrogation follow-up visits will not reveal the device type.

The physicians attending the follow-up visits and entering all patients' data into web-based CRF will be blinded to the implanted device type.

In case of an emergency with a need to reveal the type of the device, i.e. lead fracture, infection in the place of implantation, ventricular tachycardia, the site principal investigator will decide to unblind the patient. This will be documented in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of screening
* Documented non-ischemic HF with an LVEF ≤ 35
* QRS≥130ms; NYHA class II-IV
* Signed written informed consent
* NT-proBNP above 200 pg/ml

Exclusion Criteria:

* Uncorrected congenital heart disease or valve obstruction
* obstructive cardiomyopathy
* active myocarditis
* constrictive pericarditis
* untreated hypothyroidism or hyperthyroidism
* adrenal insufficiency
* active vasculitis due to collagen vascular disease
* Presence on the urgent waiting list for a heart transplant (UNOS category 1A or 1B, or equivalent)
* Patients on the non-urgent waiting list for a heart transplant (UNOS category 2 or 7, or equivalent) are eligible for inclusion in the study
* Recipient of any major organ transplant (e.g., lung, liver, heart)
* Receiving or has received cytotoxic or cytostatic chemotherapy and/or radiation therapy for treatment of a malignancy within 6 month before randomization or clinical evidence of current malignancy, with the following exceptions: basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, prostate cancer (if stable localized disease, with a life expectancy of > 2.5 years in the opinion of the investigator)
* Known to be human immunodeficiency virus positive with an expected survival of less than 5 years due to HIV
* Chronic kidney disease with glomerular filtration rate <30 ml/min
* Chronic dialysis treatment
* Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self-report
* Any condition (e.g., psychiatric illness) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Unwilling to participate

Additional information related to inclusion and exclusion criteria:

* The qualifying LVEF and NT-proBNP level has to be measured after a maximal tolerated pharmacotherapy of heart failure has been achieved.
* A non-ischemic cause of HF has to be determined by coronary angiography. Patients could be included even if they will have one or two coronary arteries with stenosis, if the extent of coronary artery disease will not be considered to be sufficient to account for the reduced LVEF. Patients with a significant coronary heart disease (CAD) will be excluded.
* Patients with an existing conventional pacemaker could be included if they will be willing to have the device changed or upgraded.
* Patients with any form of atrial fibrillation will not be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization for heart failure | 0-3 years after device implantation
  Event rate
Ventricular tachycardia | 0-3 years after device implantation
  Event rate, sustained ventricular tachycardia documentation during follow-up
Major adverse cardiac events (MACE) | 0-3 years after device implantation
  Event rate of MACE, defined as a composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death

SECONDARY OUTCOMES:
Sudden cardiac death | 0-3 years after device implantation
  Event rate of sudden cardiac death
Cardiovascular death | 0-3 years after device implantation
  Event rate of cardiovascular death
Resuscitated cardiac arrest or sustained ventricular tachycardia | 0-3 years after device implantation
  Event rate of resuscitated cardiac arrest or sustained ventricular tachycardia
Device-related complications | 0-3 years after device implantation
  Event rate of any complication requiring hospitalization
The impact in terms of overall quality of life by the SF-36 Questionnaire | 3 years after device implantation
  The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100. The lower the score the more disability. The higher the score the less disability.
The impact in terms of overall quality of life by the MacNew Questionnaire | 3 years after device implantation
  The MacNew consists of 27 items which fall into three domains: 13-item physical limitations domain scale, 14-item emotional function domain scale, 13-item social function domain scale. The maximum possible score in any domain is 7 (high QoL). The minimum is 1 (low QoL). Missing responses do not contribute to the score.

CONTACTS AND LOCATIONS:
Overall Officials: Milos Taborsky, MD, PhD, Study Director — University Hospital Olomouc
Locations (1):
- University hospital Olomouc, Olomouc, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD are to be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 6 months after the study results are published.
Access Criteria: The requests to gain access to IPD will be reviewed by National principal investigator.

REFERENCES:
- [Background] Felker GM, Thompson RE, Hare JM, Hruban RH, Clemetson DE, Howard DL, Baughman KL, Kasper EK. Underlying causes and long-term survival in patients with initially unexplained cardiomyopathy. N Engl J Med. 2000 Apr 13;342(15):1077-84. doi: 10.1056/NEJM200004133421502. PMID 10760308
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Kober L, Thune JJ, Nielsen JC, Haarbo J, Videbaek L, Korup E, Jensen G, Hildebrandt P, Steffensen FH, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Videbaek R, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S; DANISH Investigators. Defibrillator Implantation in Patients with Nonischemic Systolic Heart Failure. N Engl J Med. 2016 Sep 29;375(13):1221-30. doi: 10.1056/NEJMoa1608029. Epub 2016 Aug 27. PMID 27571011
- [Background] Bansch D, Antz M, Boczor S, Volkmer M, Tebbenjohanns J, Seidl K, Block M, Gietzen F, Berger J, Kuck KH. Primary prevention of sudden cardiac death in idiopathic dilated cardiomyopathy: the Cardiomyopathy Trial (CAT). Circulation. 2002 Mar 26;105(12):1453-8. doi: 10.1161/01.cir.0000012350.99718.ad. PMID 11914254
- [Background] Strickberger SA, Hummel JD, Bartlett TG, Frumin HI, Schuger CD, Beau SL, Bitar C, Morady F; AMIOVIRT Investigators. Amiodarone versus implantable cardioverter-defibrillator:randomized trial in patients with nonischemic dilated cardiomyopathy and asymptomatic nonsustained ventricular tachycardia--AMIOVIRT. J Am Coll Cardiol. 2003 May 21;41(10):1707-12. doi: 10.1016/s0735-1097(03)00297-3. PMID 12767651
- [Background] Kadish A, Dyer A, Daubert JP, Quigg R, Estes NA, Anderson KP, Calkins H, Hoch D, Goldberger J, Shalaby A, Sanders WE, Schaechter A, Levine JH; Defibrillators in Non-Ischemic Cardiomyopathy Treatment Evaluation (DEFINITE) Investigators. Prophylactic defibrillator implantation in patients with nonischemic dilated cardiomyopathy. N Engl J Med. 2004 May 20;350(21):2151-8. doi: 10.1056/NEJMoa033088. PMID 15152060
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Stavrakis S, Asad Z, Reynolds D. Implantable Cardioverter Defibrillators for Primary Prevention of Mortality in Patients With Nonischemic Cardiomyopathy: A Meta-Analysis of Randomized Controlled Trials. J Cardiovasc Electrophysiol. 2017 Jun;28(6):659-665. doi: 10.1111/jce.13204. Epub 2017 Apr 18. PMID 28316104
- [Background] Shen L, Jhund PS, Petrie MC, Claggett BL, Barlera S, Cleland JGF, Dargie HJ, Granger CB, Kjekshus J, Kober L, Latini R, Maggioni AP, Packer M, Pitt B, Solomon SD, Swedberg K, Tavazzi L, Wikstrand J, Zannad F, Zile MR, McMurray JJV. Declining Risk of Sudden Death in Heart Failure. N Engl J Med. 2017 Jul 6;377(1):41-51. doi: 10.1056/NEJMoa1609758. PMID 28679089
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Hawkins NM, Grubisic M, Andrade JG, Huang F, Ding L, Gao M, Bashir J. Long-term complications, reoperations and survival following cardioverter-defibrillator implant. Heart. 2018 Feb;104(3):237-243. doi: 10.1136/heartjnl-2017-311638. Epub 2017 Jul 26. PMID 28747313
- [Background] Haugaa KH, Tilz R, Boveda S, Dobreanu D, Sciaraffia E, Mansourati J, Papiashvili G, Dagres N. Implantable cardioverter defibrillator use for primary prevention in ischaemic and non-ischaemic heart disease-indications in the post-DANISH trial era: results of the European Heart Rhythm Association survey. Europace. 2017 Apr 1;19(4):660-664. doi: 10.1093/europace/eux089. PMID 28431077
- [Background] Disertori M, Mase M, Ravelli F. Myocardial fibrosis predicts ventricular tachyarrhythmias. Trends Cardiovasc Med. 2017 Jul;27(5):363-372. doi: 10.1016/j.tcm.2017.01.011. Epub 2017 Feb 2. PMID 28262437
- [Background] Gulati A, Jabbour A, Ismail TF, Guha K, Khwaja J, Raza S, Morarji K, Brown TD, Ismail NA, Dweck MR, Di Pietro E, Roughton M, Wage R, Daryani Y, O'Hanlon R, Sheppard MN, Alpendurada F, Lyon AR, Cook SA, Cowie MR, Assomull RG, Pennell DJ, Prasad SK. Association of fibrosis with mortality and sudden cardiac death in patients with nonischemic dilated cardiomyopathy. JAMA. 2013 Mar 6;309(9):896-908. doi: 10.1001/jama.2013.1363. PMID 23462786
- [Background] Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Stat Med. 1990 Dec;9(12):1447-54. doi: 10.1002/sim.4780091208. PMID 2281232
- [Background] Gart JJ, Nam J. Approximate interval estimation of the ratio of binomial parameters: a review and corrections for skewness. Biometrics. 1988 Jun;44(2):323-38. PMID 3291957
- [Background] Gart JJ, Nam JM. Approximate interval estimation of the difference in binomial parameters: correction for skewness and extension to multiple tables. Biometrics. 1990 Sep;46(3):637-43. PMID 2242407
- [Background] Kutyifa V, Geller L, Bogyi P, Zima E, Aktas MK, Ozcan EE, Becker D, Nagy VK, Kosztin A, Szilagyi S, Merkely B. Effect of cardiac resynchronization therapy with implantable cardioverter defibrillator versus cardiac resynchronization therapy with pacemaker on mortality in heart failure patients: results of a high-volume, single-centre experience. Eur J Heart Fail. 2014 Dec;16(12):1323-30. doi: 10.1002/ejhf.185. Epub 2014 Nov 7. PMID 25379962
- [Background] Barra S, Providencia R, Boveda S, Duehmke R, Narayanan K, Chow AW, Piot O, Klug D, Defaye P, Gras D, Deharo JC, Milliez P, Da Costa A, Mondoly P, Gonzalez-Panizo J, Leclercq C, Heck P, Virdee M, Sadoul N, Le Heuzey JY, Marijon E. Device complications with addition of defibrillation to cardiac resynchronisation therapy for primary prevention. Heart. 2018 Sep;104(18):1529-1535. doi: 10.1136/heartjnl-2017-312546. Epub 2018 Mar 14. PMID 29540431
- [Background] Dichtl W, Wolber T, Paoli U, Brullmann S, Stuhlinger M, Berger T, Spuller K, Strasak A, Pachinger O, Haegeli LM, Duru F, Hintringer F. Appropriate therapy but not inappropriate shocks predict survival in implantable cardioverter defibrillator patients. Clin Cardiol. 2011 Jul;34(7):433-6. doi: 10.1002/clc.20910. Epub 2011 Jun 15. PMID 21678454
- [Background] Petrie MC, Connelly DT, Gardner RS. Who needs an implantable cardioverter-defibrillator? Controversies and opportunities after DANISH. Eur J Heart Fail. 2018 Mar;20(3):413-416. doi: 10.1002/ejhf.1135. Epub 2018 Jan 12. No abstract available. PMID 29327793
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Dixon T, Lim LL, Oldridge NB. The MacNew heart disease health-related quality of life instrument: reference data for users. Qual Life Res. 2002 Mar;11(2):173-83. doi: 10.1023/a:1015005109731. PMID 12018740
- [Derived] Taborsky M, Skala T, Aiglova R, Fedorco M, Kautzner J, Jandik T, Vancura V, Linhart A, Valek M, Novak M, Kala P, Polasek R, Roubicek T, Schee A, Hindricks G, Dagres N, Hatala R, Jarkovsky J. Cardiac Resynchronization and Defibrillator Therapy (CRT-D) or CRT Alone (CRT-P) in patients with dilated cardiomyopathy and heart failure without late gadolinium enhancement (LGE) cardiac magnetic resonance imaging (CMRI) high-risk markers - CRT-REALITY study - Study design and rationale. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 May;166(2):173-179. doi: 10.5507/bp.2021.015. Epub 2021 Mar 12. PMID 33724264